CLINICAL TRIAL: NCT05182762
Title: Measuring Quality in Colorectal Cancer Surgery in Low- and Middle-income Countries: the Clavien-Dindo Classification in a Sri Lankan Cohort
Brief Title: Measuring Quality in Colorectal Cancer Surgery in Low- and Middle-income Countries
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, David Ljungman, Consultant surgeon, Sahlgrenska University Hospital
Other Study IDs: MO/PLEC/2020:822
Record Dates: First submitted 2021-12-08; First posted 2022-01-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Colorectal Cancer; Postoperative Complications; Surgical Complication; Non-communicable Disease
Keywords: Colorectal cancer; Sri Lanka; Clavien-Dindo Classification; Postoperative complications; Surgical quality
MeSH Terms: conditions — Colorectal Neoplasms; Postoperative Complications; Noncommunicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To test the applicability of the Clavien-Dindo Classification (CDC) in an LMIC setting and to compare the prevalence and severity of complications in patients <60 and ≥60 years of age a retrospective medical records review is used.

DETAILED DESCRIPTION:
Background: Colorectal cancer (CRC) is increasing in Low- and Middle-Income Countries (LMIC) as part of the ongoing epidemiological transition. Surgery is the main treatment and the global health agenda is increasingly putting focus on improving the safety and quality of surgical care in low-resource settings. The current systems for measuring surgical quality are mainly customized for high-income countries.

Aim: To test the applicability of the Clavien-Dindo Classification (CDC) in an LMIC setting. Additionally, to compare the prevalence and severity of complications in patients <60 and ≥60 years of age.

Material and methods: Retrospective medical records review for postoperative complications and severity grading using the CDC.

ELIGIBILITY:
Inclusion Criteria:

* Patients who has gone through colorectal cancer resection.
* Surgery performed at Colombo South Teaching Hospital in Colombo, Sri Lanka.

Exclusion Criteria:

* Reason for resection other than colorectal cancer.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 100 consecutive patients retrospectively collected from the medical journals at Colombo South Teaching Hospital in Colombo, Sri Lanka.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Clavien-Dindo Grade | February 2020 to March 2020
  Postoperative complications graded by the Clavien-Dindo Classification.

SECONDARY OUTCOMES:
Age comparison | February 2020 to March 2020
  Comparison of prevalence and severity of complications between patients <60 and ≥60 years of age.

CONTACTS AND LOCATIONS:
Overall Officials: David Ljungman, MD PhD, Study Director — Dep. of Surgery, Institute of Clinical Sciences, Sahlgrenska Academy, University of Gothenburg..; Stina Lindholm, MD, Principal Investigator — Sahlgrenska Academy, University of Gothenburg.; Sofia Lindskogen, MD, Principal Investigator — Sahlgrenska Academy, University of Gothenburg.; Göran Kurlberg, Asoc prof, Study Director — Dep. of Surgery, Institute of Clinical Sciences, Sahlgrenska Academy, University of Gothenburg.; Bawantha Gamage, MD, Study Director — Dep. of Surgery, Colombo South Teaching Hospital, University of Sri Jayewardenepura.
Locations (1):
- University of Gothenburg, Sahlgrenska Academy, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT05182762/Prot_SAP_ICF_000.pdf